CLINICAL TRIAL: NCT06863428
Title: Concordance Between an App-based Range of Motion Measurement and Standard Goniometer.
Brief Title: Mymobility Knee ROM
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2024-28TDS
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Knee Range of Motion
Keywords: mymobility; range of motion; goniometer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: This group will have their knee range of motion measured three times. Once with the mymobility app, and twice using a goniometer by two separate assessors. Each assessor will be blinded to the other assessor's measurements.

SUMMARY:
This prospective study aims to evaluate the agreement, also referred as concordance, of the mymobilty knee ROM with a clinician's assessment of knee ROM via goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years of age
* Patient is willing and able to provide written Informed Consent by signing and dating the IRB-approved Informed Consent form

Exclusion Criteria:

* The patient is currently participating in any other study that would hinder the assessor's ability to measure knee ROM
* Complex primary knee pathology with significant restrictions on the range of motion per surgeon discretion
* Patient is pregnant or considered a member of a protected population (e.g. prisoner, mentally incompetent, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a minimum of 41 patients who meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Active knee flexion | Day 1 (Single Visit)
  Patients will be asked to sit in a chair to measure full active knee flexion.
Active knee extension | Day 1 (Single Visit)
  Patients will be asked to sit in a chair to measure full active knee extension.
Passive knee extension with overpressure | Day 1 (Single Visit)
  Patients will be asked to sit in a chair to measure full passive knee extension while applying overpressure on their knee with their hands.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (1):
- Center for Advanced Orthopedics and Sports Medicine, Auburn Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No